CLINICAL TRIAL: NCT02587455
Title: Phase I Dose Escalation of pAlliative Radiotherapy With Anti-PD1 Antibody Pembrolizumab in Thoracic Tumours
Brief Title: Pembrolizumab and Palliative Radiotherapy in Lung
Acronym: PEAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Institute of Cancer Research, United Kingdom (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCR 4282
Record Dates: First submitted 2015-10-13; First posted 2015-10-27 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Thoracic Tumours
Keywords: Non-small cell carcinoma
MeSH Terms: interventions — pembrolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose Radiotherapy Arm (Experimental): Pembrolizumab and radiotherapy
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy
- High Dose Radiotherapy Arm (Experimental): Pembrolizumab and radiotherapy
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab - Trial Treatment
  Other Names: MK-3475/pembrolizumab (KEYTRUDA®)
Radiation: Radiotherapy — Radiotherapy - Standard Treatment

SUMMARY:
Lung cancer is the second most common cancer in the UK with around 43,500 new patients diagnosed each year. About 69% of patients are diagnosed with advanced stage disease and at present these patients would be expected to survive for less than 12 months. These statistics therefore show the need for the development of new effective drugs in the treatment of advanced Lung cancer.

Recent trial results have shown the efficacy of immunotherapy in treating several types of tumours including lung cancer. These tumours are known to express a high level of a glycoprotein called PDL1 which is a component of the PD1 pathway. In cancer the PD1 pathway can be hijacked by tumours leading to the immune system being suppressed. The aim of the new drug Pembrolizumab is to restart the PD1 pathway and use the immune system to help fight the cancer cells. Radiotherapy has also been shown to cause cancer to increase production of the proteins that can block the immune system. Therefore it has been proposed that combine of new immunotherapy agent such as pembrolizumab and radiotherapy in the treatment of lung cancer will allow more cancer cells to be killed through the immune system.

The purpose of this study is to see if pembrolizumab can safety be combined with standard palliative radiotherapy in patients with lung cancer. In addition once the patients have completed their course of radiotherapy they will remain on pembrolizumab alone and the study will look at how well this treatment regimen can control the growth of the cancer.

DETAILED DESCRIPTION:
1. Risk and burden for patients

   Patients in the first part of this study have cancer that is no longer responding to standard anticancer drug treatments.The phase 1 nature of this study means that the trial intervention may not have any additional benefit for patients who take part in the study.

   The study itself carries a number of potential burdens:
   * Study drug and radiotherapy:

   Although the study drug safety effects have previously been assessed in NSCLC the side effects caused by the addition of radiotherapy is unconfirmed. These risks will be managed as much as possible by cautious dose escalation: as with all phase 1 studies, the data from each cohort will be reviewed by a safety review committee before deciding whether to increase the dose for subsequent cohorts.

   Participants will be reviewed regularly by experienced clinicians while having the study treatment. Comprehensive assessments for safety will be carried out.
   * Burden of frequent hospital visits and tests:

   Participants in this study must attend hospital frequently, particularly at the start of the study, for safety reasons to check for any toxicity of the study treatment. Blood tests, clinical examination, urine tests, haematology, bio chemistry and lung function tests are part of the safety assessment. Additionally, for research purposes some participants may be asked to have additional blood taken, these will not be mandatory for entry into the study.
2. Recruitment

Participants will be offered information about this study by their clinical teams if they are considered to meet the entry criteria (with regard to advanced disease without therapeutic option, suitable performance status) and express interest in taking part in an experimental study. It will be made clear that the study is experimental in nature and that there will not necessarily be a therapeutic benefit from taking part in the study. It will also be made clear that, should patients decide not to take part their future care will not be affected. Patients will be given sufficient time and information to make an informed decision about entering the trial, all patients entering the trial will give written informed consent.

4. Confidentiality

Patients will be linked to a unique identifier the code for which will be held on a password protected database held only by the study team. This study will run at the Royal Marsden Hospital Only. Research blood and tumour data will be analysed by a team at the Institute of cancer Research. Sample processing will take place using the trial ID only. No other patient identifiable information will be available on study samples. Investigators will have access to patient identifiable information on password protected NHS hospital notes and databases only.

5. Conflict of Interest

Patients may be recruited to the study by those involved in their prior clinical care. The investigators do not expect conflict of interest between research and healthcare duties for a number of reasons: patients must give their full informed consent before entering the study, specifically regarding the unknown efficacy of the study drug. Those patients who do not continue in the study will maintain a relationship with the clinical team if required for symptom control. At the end of the study, patients will be able to access the results if they wish, through the Royal Marsden Website. They will also be sent a written summary of the results if they indicate this.

6. Use of tissue samples in future research

If participants give their consent, any leftover blood or tissue samples which are not required for this study will be stored for future unspecified research in line with the human tissue act regulations. Access and use of samples for research purposes will require appropriate ethical approval. Future researchers will not be able to identify individual patients from their biobank data, demographic and clinical information will be available.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Have measurable disease based on RECIST 1.1.
3. Histologically verified NSCLC including squamous cell carcinoma, adenocarcinoma, adenosquamous or large cell anaplastic carcinoma; requiring palliative radiotherapy for which no curative therapy exists will be recruited into the trial.
4. Patients are permitted to have extrathoracic disease which will not be encompassed in the radiotherapy field. This disease will be assessed for abscopal response
5. Ability to tolerate a course of palliative radiotherapy to the lung.
6. Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumour lesion.
7. Have a performance status of 0-2 on the ECOG Performance Scale.
8. Demonstrate adequate organ function, all screening labs should be performed within 10 days of confirmation of eligibility.
9. Patient's lung function tests at baseline should have an FEV1 > 0.8L or > 30%.
10. See protocol section.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Previous radiotherapy to the lung
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   Note: Patients with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require the use of bronchodilators or local steroid injections would not be excluded from the study. Patients with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
9. Has evidence of interstitial lung disease or active, noninfectious pneumonitis.
10. Has received prior therapy with an antiPD1, antiPDL1, antiPDL2, antiCD137, or anti Cytotoxic T-lymphocyte associated antigen4 (CTLA4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways).
11. See protocol section.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Toxicity rate of DLTs assessed by CTCAEv4 | two months after the last fraction of RT has been administered
Maximum tolerated dose (MTD) of pembrolizumab that can be safely combined with radiotherapy (RT) in the absence of dose limiting toxicity (DLT) assessed by CTCAEv4 | up to 24 months

SECONDARY OUTCOMES:
Progression free survival rates will be calculated at 6 and 12 months, respectively | 6 and 12 months
Overall survival rates will be calculated at 6 and 12 months, respectively | 6 and 12 months
Progression free survival rates will be calculated at 6 and 12 months for PDL-1 strong patients, respectively | 6 and 12 months
Overall survival rates will be calculated at 6 and 12 months for PDL-1 strong patients, respectively | 6 and 12 months
Duration of clinical benefit, as assessed by RECIST v1.1 | 6 months and 1 year
Compare response rates, as assessed by RECIST v1.1, between squamous and non-squamous histological sub-types | 6 months and 1 year

OTHER OUTCOMES:
Assessing individual lesion response (CR/PR/PD/SD) determined by RECIST v1.1 to evaluate the abscopal effect between pembrolizumab and RT | cycle 2 (week 8/9) and cycle 5 (week 17/18)
Identify biomarkers and correlate with clinical benefit, as defined by RECIST v1.1 | through study completion (24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Merina Ahmed, Study Director — Consultant Clinical Oncologist
Locations (2):
- United Kingdom (2):
  - NIHR Biomedical Research Centre at RM and ICR (https://www.cancerbrc.org/), London
  - NIHR Biomedical Research Centre at RM and ICR (https://www.cancerbrc.org/), Sutton